CLINICAL TRIAL: NCT02790931
Title: Effects of Foot Muscle Strengthening in Daily Activity, Biomechanics and Functionality of Foot and Ankle in Diabetic Polyneuropathy Patients: a Randomized Controlled Trial
Brief Title: Effects of Foot Muscle Strengthening in Daily Activity in Diabetic Neuropathic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Isabel de Camargo Neves Sacco, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LaBiMPH
Record Dates: First submitted 2016-05-25; First posted 2016-06-06 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Neuropathies
Keywords: diabetic foot; therapeutic exercises; foot; preventive care; rehabilitation; Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Patients will receive a physical therapy intervention in groups twice/wk, and using a software twice/ wk for 3 months.
  Interventions: Other: Intervention Group
- Control Group (No Intervention): Patients will not receive any exercise treatment, will not have acess to the software, but they will keep their recommended clinical treatment.

INTERVENTIONS:
Other: Intervention Group — Patients will receive a physical therapy intervention in groups twice/wk, and using a software twice/ wk for 3 months, for foot and ankle strengthening, stretching and functional training. They must continue to exercise at home twice a week with the software supervision for one year.
  Other Names: Foot and ankle kinesiotherapy
  Arms: Intervention Group

SUMMARY:
The main objective of this trial is to investigate the effects of foot muscle strengthening in daily activity of patients with diabetic neuropathy.

DETAILED DESCRIPTION:
A randomized controlled trial will be performed with 77 patients with diabetic neuropathy. The participants will be randomly assigned into either a control group (recommended foot care by international consensus with no exercises) or an intervention group which will receive 12-week physical therapy exercises, twice a week, under the supervision of a physiotherapist, and twice a week being remotely supervised by a software at home. Every exercise has its own progression depending on the subjects' execution, increasing in intensity and difficulty.

The subjects will be evaluated in 5 different moments (Baseline, 6 weeks, 12 weeks, 24 weeks and 1 year follow-up)

The hypothesis of this study is that the intervention group will increase daily activity levels, increase self-selected and rapid walking speed, reduce the incidence of plantar ulcers, increase foot health and functionality, improve symptoms, increase tactile and vibration sensitivity, increased passive range of motion, improved quality of life, increased isometric strength of the feet and production of beneficial biomechanical changes during walking compared to the control group after 12 weeks of intervention and follow-up year.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or 2
* Moderate or severe polyneuropathy confirmed with the fuzzy software
* Ability to walk independently in the laboratory
* Accessibility to electronic devices
* Loss of at least 4 degrees of ankle range of motion
* Loss of at least 1 degree of force in the clinical scale of the plantar interosseous or lumbrical muscles

Exclusion Criteria:

* Ulceration not healed for at least 6 months
* Hallux amputation or total amputation of the foot
* Receiving any physiotherapy intervention or offloading devices
* Neurological or orthopedic impairments
* Major vascular complications
* Severe retinopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-08; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel CN Sacco, PhD, Principal Investigator — Associate Professor at São Paulo University
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monteiro RL, Ferreira JSSP, Silva EQ, Cruvinel-Junior RH, Verissimo JL, Bus SA, Sacco ICN. Foot-ankle therapeutic exercise program can improve gait speed in people with diabetic neuropathy: a randomized controlled trial. Sci Rep. 2022 May 9;12(1):7561. doi: 10.1038/s41598-022-11745-0. PMID 35534614
- [Derived] Monteiro RL, Sartor CD, Ferreira JSSP, Dantas MGB, Bus SA, Sacco ICN. Protocol for evaluating the effects of a foot-ankle therapeutic exercise program on daily activity, foot-ankle functionality, and biomechanics in people with diabetic polyneuropathy: a randomized controlled trial. BMC Musculoskelet Disord. 2018 Nov 14;19(1):400. doi: 10.1186/s12891-018-2323-0. PMID 30428863
- See also: Laboratory of Biomechanics of Human Movement and Posture website — http://www.usp.br/labimph
- See also: University of Sao Paulo website — http://www.usp.br/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was enrolled 78 participants (1 more than the protocol) because the main research intended to keep the number of participants in each group equal.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 39 | 39
Completed | 15 | 19
Not Completed | 24 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.7) | 60.1 (8.9) | 60.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 39 | 39 | 78
Daily physical activity [Mean (Standard Deviation); unit: Total Steps per week] | 8.092 (4.230) | 7.641 (4.087) | 7.866 (4158)
Fast gait speed [Mean (Standard Deviation); unit: m/s] | 1.5 (0.2) | 1.5 (0.3) | 1.5 (0.25)
Self-selected gait speed [Mean (Standard Deviation); unit: m/s] | 1.1 (0.2) | 1.0 (0.1) | 1.0 (0.15)
Height [Mean (Standard Deviation); unit: m] | 1.6 (0.08) | 1.6 (0.09) | 1.6 (0.08)
Body mass [Mean (Standard Deviation); unit: kg] | 77.3 (14.0) | 80.8 (16.4) | 79 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Daily Physical Activity
Description: Calculate the number of steps per week
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: number of steps per week
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 22 | 12
number of steps per week | 8744 (810) | 7373 (1010)

2. Primary Outcome: Self Selected Gait Speed
Description: self selected gait speed shod walking velocity in a walkway
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 24 | 17
m/s | 1.06 (0.04) | 1.00 (0.04)

3. Primary Outcome: Fast Gait Speed
Description: Fast gait speed shod walking velocity in a walkway
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 24 | 17
m/s | 1.68 (0.06) | 1.49 (0.06)

4. Secondary Outcome: Risk Classification of Plantar Ulceration
Description: Score of the classification of the plantar ulcer risk (IWG diabetic foot)
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Foot Health and Functionality
Description: Score of the Foot Health Status questionnaire - BRAZIL
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Foot Strength
Description: Hallux and lesser toes force measured by a pressure plate
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Foot and Ankle Kinematics During Gait
Description: Foot joints and plantar arch motion, ankle range of motion, and maximum ankle extension and flexion during gait
Time Frame: baseline, 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Ankle and Knee Joint Moments and Power During Gait
Description: Peak joint moment and eccentric and concentric power by inverse dynamic calculations
Time Frame: baseline, 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Plantar Ulcers
Description: New cases of foot plantar ulcers
Time Frame: 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Tactile Sensitivity
Description: Evaluation of the tactile sensitivity of four plantar areas with 10g monofilament
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Vibration Sensitivity
Description: Evaluation of the vibration sensitivity with tuning fork
Time Frame: 12 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Neuropathy Symptoms
Description: Score of the Michigan Neuropathy Screening Instrument questionnaire Michigan Neuropathy Screening Instrument (MNSI)
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Range of Motion
Description: Manual goniometry of the range of motion of flexion and extension of the metatarsophalangeal joint of the hallux and ankle.
Time Frame: 12 weeks
Reporting Status: Not Posted

14. Secondary Outcome: EQ-5D Score
Description: EQ-5D score of the quality of life of the patient
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the intervention period (aproximately 12 weeks)
Description: There was no serious adverse and all-cause mortality in the control and in the intervention groups.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT02790931/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02790931/ICF_001.pdf